CLINICAL TRIAL: NCT06072430
Title: A Phase III, Open Label, Randomized, Controlled Study of VBI-S in the Treatment of Hypovolemia in Patients With Septic Shock
Brief Title: A Phase III, Open Label, Randomized, Controlled Study of VBI-S in the Treatment of Hypovolemia in Patients With Septic Shock (VBI-S-02)
Acronym: VBI-S-02
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Vivacelle Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VBI-S-02
Record Dates: First submitted 2023-09-14; First posted 2023-10-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Septic Shock; Sepsis; Hypovolemia
MeSH Terms: conditions — Shock, Septic; Sepsis; Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- VBI-S (Experimental): Treatment with VBI-S
  Interventions: Drug: VBI-S

INTERVENTIONS:
Drug: VBI-S — VBI-S is made of small particles of specific lipids called micelles and liposomes for the treatment of hypotension.

SUMMARY:
This study is being conducted to evaluate the safety and effectiveness of VBI-S in elevating the blood pressure of septic shock patients with absolute or relative hypovolemia.

DETAILED DESCRIPTION:
PURPOSE OF THE STUDY This study is being conducted to evaluate the safety and effectiveness of VBI-S in elevating the blood pressure of septic shock patients with absolute or relative hypovolemia.

STUDY TREATMENT Sepsis is a serious condition resulting from the presence of harmful microorganisms in the blood or other tissues and the body's response to their presence, leading to the malfunctioning of various organs. When hypotension due to sepsis cannot be reversed with the infusion of fluids the patient is in a state of septic shock. Septic shock is therefore an acute medical emergency and delayed therapy can lead to organ injury. VBI-S is intended to raise blood pressure in patients with septic shock.

Randomization and blinding: This is a randomized, controlled, open-label study and blinding is not applicable to this study.

Data Safety Monitoring Board: A Data Safety Monitoring Board (DSMB) will review the study data.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female at least 18 years of age.
2. Evidence of bacterial infection demonstrated by positive blood culture and/or a known source of infection and/or an elevated procalcitonin of ≥ 2 ng/ml.
3. Patient has a mean blood pressure < 65 mmHg that is unresponsive to fluids currently available on the market.
4. Sequential Organ Failure Assessment (SOFA) score ≥ 5
5. Sepsis diagnosis: The presence of infection which can be proven or suspected by 2 or more of the following criteria:

   * Lactate > 2 mmol/L
   * Fever > 38.3°C, or 101°F
   * Hypothermia < 36°C core temperature (<96.8°F)
   * Heart rate > 90
   * Tachypnea (respiratory rate ≥ 20/min)
   * White blood cell count >12,000 or less than 4,000, or with >10% "bands" (immature forms)
   * Elevated procalcitonin in serum (≥ 2ng/ml)
   * Arterial hypoxemia (PaO2/FiO2 < 300)
   * Creatinine increase > 0.5 mg/dL since hospital admission
   * INR > 1.5 or aPTT > 60 seconds
6. Documented dysregulated host response to an infection as indicated by an increase in SOFA score by ≥ 2 points after an infection per the SEPSIS 3 guideline.
7. Receiving vasopressors to maintain the target MAP of 65 mmHg.

Exclusion Criteria:

1. Patients with a ventricular assist device
2. Acute coronary syndrome
3. Pregnant
4. Acute bronchospasm
5. Acute Mesenteric ischemia
6. Emergency major surgery
7. Diagnosis of acute Hepatitis B or C.
8. Hematologic or coagulation disorders including thrombocytopenia (platelet count <50,000) and associated with hemodynamically significant active bleeding that causes a decrease in blood pressure.
9. White blood cell count of < 1000 mm3
10. Current participation or participation in another experimental or device study within the last 30 days before the start of this study. Patient may be included if on other drugs are for COVID-19.
11. Patients with a known allergy to soybeans or eggs
12. Patient is hypervolemic with assessment by physician or physician extender ultrasound 12 hours before infusion of VBI-S if hypervolemia is suspected.
13. Patient expected to expire within 12 hours.
14. Patients with disturbances in normal fat metabolism such as pathologic hyperlipemia, lipid nephrosis, or acute pancreatitis with hyperlipidemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Elevation in Average Mean Arterial Pressure | 12 months
  The primary endpoint is defined as an elevation in average mean arterial pressure by at least 10 mmHg from baseline within 3 hours of initiation of study treatment on Day 1

SECONDARY OUTCOMES:
Dose of Pressor Drugs | 12 months
  The number of patients in whom the dose of pressor drugs could be decreased after infusion of VBI-S to maintain a mean arterial pressure of 60-65 mmHg.
Sequential Organ Failure Assessment (SOFA) Score | 12 months
  Change in Sequential Organ Failure Assessment (SOFA) Score on a scale of 0 to 24. A higher score indicates a worse outcome.
Ratio of Arterial Partial Pressure of Oxygen/Fraction of Inspired Oxygen | 12 months
  Change in ratio of partial pressure of oxygen in arterial blood/Fraction of inspired oxygen (P/F ratio).
Arterial Oxygen Saturation | 12 months
  Change in arterial oxygen saturation.
Partial Pressure of Oxygen | 12 months
  Change in partial pressure of oxygen.
Serum Procalcitonin | 12 months
  Change in serum procalcitonin
Serum Creatinine | 12 months
  Change serum creatinine
Post-treatment Survival | 12 months
  Change in post-treatment survival

OTHER OUTCOMES:
Adverse Drug Reactions | 12 months
  The number and proportion (%) of patients with treatment-emergent adverse drug reactions.

CONTACTS AND LOCATIONS:
Overall Officials: Cuthbert O Simpkins, MD, FACS, Principal Investigator — Vivacelle Bio
Locations (6):
- United States (6):
  - Dignity Health Chandler Regional Medical Center, Chandler, Arizona
  - Memorial Health University Medical Center, Savannah, Georgia
  - University Health, Kansas City, Missouri
  - Bryan Medical Center, Lincoln, Nebraska
  - Novant Healthcare, Winston-Salem, North Carolina
  - Oregon Health & Science University (OHSU), Portland, Oregon

IPD SHARING:
Plan to Share IPD: No